CLINICAL TRIAL: NCT06403280
Title: The Effect of Alcohol on Common Tremor Syndromes - A Prospective Double-blind Randomised Cross-over (Alcohol, Placebo) Study
Brief Title: The Effect of Alcohol on Common Tremor Syndromes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EK 35-415 ex 22/23
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Essential Tremor; Dystonia; Parkinson Disease
Keywords: accelerometry; alcohol responsiveness
MeSH Terms: conditions — Essential Tremor; Dystonia; Parkinson Disease | interventions — Alcoholic Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Day (Experimental): Participants will receive vodka with rum flavored orange juice with a target blood alcohol of 0.4 ‰ 30 minutes after alcohol consumption. The required amount of vodka will be calculated with the Widmark formula.
  Interventions: Dietary Supplement: Alcoholic drink
- Placebo Day (Placebo Comparator): Participants will receive a non-alcoholic rum flavored orange juice.
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Alcoholic drink — Participants will receive vodka with rum flavored orange juice with a target blood alcohol of 0.4 ‰ 30 minutes after alcohol consumption. The required amount of vodka will be calculated with the Widmark formula.
  Arms: Interventional Day
Dietary Supplement: Placebo drink — Participants will receive a non-alcoholic rum flavored orange juice.
  Arms: Placebo Day

SUMMARY:
The aim of this interventional study is to compare the response to alcohol in patients with essential tremor (ET), essential tremor plus (ETplus), dystonic tremor (DT), tremor associated with dystonia (TaD) and tremor in Parkinson´s disease (PD). The main question to be answered is:

• Is there a difference in the objective alcohol responsiveness of patients with ET, DT, TaD and PD?

Participants will receive either vodka with rum-flavoured orange juice with a target blood alcohol of 0.4 ‰ or a non-alcoholic rum-flavoured orange juice (vice versa on the second study day). Before and 30, 60 an 120 minutes after the study drink the participants will undergo a clinical examination of the tremor and accelerometry will be performed.

Researchers will compare alcohol and placebo in a randomized cross over way to see if the effect of alcohol on tremor exceeds the placebo effect.

DETAILED DESCRIPTION:
The researchers will include 45 patients (9 each) with essential tremor (ET), essential tremor plus (ETplus), dystonic tremor (DT), tremor associated with dystonia (DaT) or tremor in Parkinson´s disease (PD) from the Movement Disorders Outpatients Clinic of the Medical University of Graz.

Participants will be asked to stop any tremor influencing medication and alcohol intake 24 hours before testing. 4 hours before testing the participants should not eat or drink anything. The participants will be asked to bring an accompanying person and are not allowed to drive at the day of the study visit.

Each participant will be examined at two different days (intervention and placebo day) with at least one day in between. During the study participation the tremor influencing medication should not be changed. The study design is a randomized cross sectional design where each participant receives either alcohol or placebo and vice versa on the second study day. The participants will be asked to finish the study drink within 15 minutes.

Interventional day:

Participants will receive vodka with rum flavored orange juice with a target blood alcohol of 0.4 ‰ 30 minutes after alcohol consumption. The required amount of vodka will be calculated with the Widmark formula.

Placebo day:

Participants will receive non-alcoholic rum flavored orange juice.

Baseline examinations:

* Questionnaire (only on the first study visit): demographics, disease duration, onset of disease, alcohol drinking habits and noticed effects of alcohol on tremor
* Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
* The Essential Tremor Ranking Scale (TETRAS)
* The Burke-Fahn-Marsden (BFM) Dystonia Rating Scale
* Placement of an indwelling venous cannula in a cubital fossa vein (for repeated blood alcohol measurements)
* Accelerometry: The participants will sit in a chair with a triaxial accelerometer transducer attached to the dorsal surface of the middle phalanx of the index finger. Each position will be recorded 30 seconds.

Recorded positions:

1. rest position: arms relaxed and hands hanging freely from the arm rest
2. posture position: arms / wrists outstretched at shoulder level

Examinations 30 minutes after the intervention (study drink):

* TETRAS Performance Subscale
* MDS-UPDRS motor examination (part III)
* BFM scale
* Accelerometry
* Evaluation of possible side effects

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD, DT, TaD, ET or ETplus based on clinical diagnostic criteria
* tremor in upper extremities
* accompanying person for both study visits

Exclusion Criteria:

* persons that are not willing to abstain from driving at both study days
* patients with diseases prohibiting alcohol ingestion
* patients with a history of alcohol abuse
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the Total Tremor Power measured by accelerometry | 30 minutes after each study drink. Duration of measurement: 5 minutes.
  The the total tremor power (TP) of the spectra between 1 and 30 Hz for each axis will be used. The square root of the sum of the squares of the TP of each accelerometer axis will be calculated. This will be the Change of the Total Tremor Power and will serve as a surrogate for tremor amplitude.

SECONDARY OUTCOMES:
Change from baseline in TETRAS-P | 30 minutes after each study drink. Duration of measurement: 3 minutes.
  Change in The Essential Tremor Rating Scale - Performance Subscale (TETRAS-P) before and after the intervention will be used as clinical parameter of tremor severity in patients with essential tremor, dystonic tremor and tremor associated with dystonia. The TETRAS-P Scale is a 16 item scale with a possible score range between 0 (=no tremor) and 64 points (=worst tremor).
Change from baseline in UPDRS III | 30 minutes after each study drink. Duration of measurement: 5 minutes.
  The change of the motor examination of the Movement Disorder Society-Unified Parkinson´s Disease Rating Scale (part 3) will be used as clinical parameter for tremor and changes in motor examination in patients with Parkinson´s Disease. The UPDRS III is a 32-items scale with a possible score range between 0 (=no motor symptoms) and 128 points (=worst result).
Change from baseline in Visual Analogue Scale (VAS) | 30 minutes after each study drink. Duration of measurement: 1 minute.
  The change in the Visual Analogue Scale (VAS) is be used to assess the subjective tremor severity. The VAS ranges from 0 to 10, with higher values indicating worse subjective tremor.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schwingenschuh, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No